CLINICAL TRIAL: NCT00245609
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Trial Of The Anxiolytic Efficacy Of Pregabalin And Alprazolam IR In Subjects With Anxiety Prior To Dental Procedure
Brief Title: Trial of Pregabalin, Alprazolam, and Placebo in Subjects With Anxiety Prior to Dental Procedure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081072
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2008-03

CONDITIONS: Dental Anxiety
MeSH Terms: interventions — Pregabalin; Alprazolam

INTERVENTIONS:
Drug: Pregabalin
Drug: Alprazolam
Drug: Placebo

SUMMARY:
The primary purpose of the trial is to assess how effective pregabalin, alprazolam, and placebo are at reducing anxiety levels of subjects who take a dose of these treatments 4 hours before a scheduled dental procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients 18 years of age or older who score 12 points or more on the Dental Anxiety Scale at screening and baseline evaluations and have a scheduled appointment for an elective dental procedure.

Exclusion Criteria:

* Current diagnosis of any of the DSM-IV anxiety disorders.
* Current diagnosis of major depressive disorder, dysthymia, schizophrenia or any other psychotic disorder, bipolar disorder, and eating disorders as assessed by the M.I.N.I. at screening, or current diagnosis of delirium, dementia, or body dysmorphic disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2006-01; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint on the Visual Analogue Scale for Anxiety.

SECONDARY OUTCOMES:
The changes from baseline to endpoint, and changes from baseline to each rating timepoint differ among the three treatment groups for the VAS-Anxiety, VAS-Sedation, Time to Onset of Activity Scales scores, and, Dental Anxiety scales.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Germany (6):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Tübingen
- United Kingdom (3):
  - Pfizer Investigational Site, Manchester, Greater Manchester
  - Pfizer Investigational Site, Leeds, West Yorkshire
  - Pfizer Investigational Site, Sheffield

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081072&StudyName=Trial+of+pregabalin%2C+alprazolam%2C+and+placebo+in+subjects+with+anxiety+prior+to+dental+procedure